CLINICAL TRIAL: NCT00217308
Title: Effect of Probiotic Lactobacilli on Vaginal Flora of Pregnant Women at High Risk for Preterm Delivery
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Tightly defined inclusion criteria were making recruitment very slow.
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Alan Bocking, Clinician Scientist, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-0169-A
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Premature Birth; Bacterial Vaginosis
MeSH Terms: conditions — Premature Birth; Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus (Experimental)
  Interventions: Drug: Lactobacilli GR-1 and RC-14
- Placebo capsules (Placebo Comparator)
  Interventions: Drug: Lactobacilli GR-1 and RC-14

INTERVENTIONS:
Drug: Lactobacilli GR-1 and RC-14 — Probiotic Lactobacilli will be compared to placebo

SUMMARY:
Purpose of the study is to determine the effect of probiotic lactobacilli on the vaginal flora and cytokine profile during pregnancy, and the incidence of preterm labour in women at high risk for preterm birth.

DETAILED DESCRIPTION:
Preterm labour involves multiple causes - one of the most significant factors being a prior history of preterm birth. Infection is another major cause of preterm labour (PTL) and is estimated to cause up to 30% of PTL. Bacterial Vaginosis (BV) is an alteration in the endogenous vaginal microflora preceded by a decreased presence of Lactobacilli species and increased growth of gardnerella and other pathogens. BV is a strong risk factor for PTL, and is associated with a 40% increased risk in some populations. Initial studies suggested that the treatment of BV with antibiotics could decrease the incidence of PTL, but this has not been confirmed by randomized trials. There is substantial evidence that the "normal" lactobacillus dominated urogenital microflora play an important role in maintenance of a healthy urinary and reproductive tract.

One hundred and sixty (160) women at high risk for PTL, based on a prior history of preterm birth, will be approached at their first antenatal visit to participate. Recruitment of 54 patients with symptomatic or asymptomatic BV (based on Nugent Scoring). Women with documented BV will be randomized to either treatment with lactobacilli preparation (n=27) or placebo (n=27). Women with symptomatic BV will be treated with oral Metronidazole prior to starting the lactobacilli or placebo. None of the subjects, researchers or clinical staff will know which preparation each woman receives.

This study will be the first to examine the ability of lactobacilli preparations to maintain a normal vaginal flora in pregnant women. In addition, the results will potentially serve as the basis for a multi-centre RCT to determine efficacy of this treatment in preventing preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with previous incidence of preterm labour
* otherwise healthy
* over 18 years of age
* able to provide informed consent
* less than or equal to 16 weeks gestation
* singleton pregnancy
* normal uterine cavity

Exclusion Criteria:

* significant medical complications (preeclampsia, thrombophilia, hypertension)
* multiple pregnancy
* less than 18 years of age
* patients receiving antibiotics or other antimicrobial therapies at time of recruitment
* fetal complications such as intrauterine growth restriction or other abnormalities
* diabetes
* documented need for cervical cerclage
* patient enrolled in other clinical trials

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-02 (Actual); Primary Completion 2007-07 (Estimated); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Determination if restoration of a normal vaginal flora through the use of probiotics reduces the incidence of PTB. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alan Bocking, MD, FRCSC, Principal Investigator — Chief, Department of Obstetrics and Gynaecology, Mount Sinai Hospital
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No